CLINICAL TRIAL: NCT00943072
Title: A Randomized, Double Masked, Controlled Phase 3 Study of the Efficacy, Safety, and Tolerability of Repeated Intravitreal Administration of Vascular Endothelial Growth Factor Trap-Eye in Subjects With Macular Edema Secondary to Central Retinal Vein Occlusion
Brief Title: Vascular Endothelial Growth Factor (VEGF) Trap-Eye: Investigation of Efficacy and Safety in Central Retinal Vein Occlusion (CRVO)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VGFT-OD-0819
Record Dates: First submitted 2009-07-10; First posted 2009-07-21 (Estimated); Results first posted 2013-05-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-04

CONDITIONS: Macular Edema Secondary to Central Retinal Vein Occlusion
Keywords: Macular edema; Retinal vein occlusion; CRVO; VEGF Trap-Eye; best-corrected visual acuity; Regeneron; COPERNICUS
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — aflibercept; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VEGF Trap-Eye (Experimental): Monthly IVT injection of VEGF Trap-Eye 2.0 mg until Week 24 Primary Endpoint
  Interventions: Biological: VEGF Trap-Eye 2.0mg
- Sham (Sham Comparator): Monthly Sham IVT injection until Week 24 Primary Endpoint
  Interventions: Drug: Sham

INTERVENTIONS:
Biological: VEGF Trap-Eye 2.0mg — Monthly intravitreal injection out to the Week 24 Primary endpoint
  Arms: VEGF Trap-Eye
Drug: Sham — Monthly sham intravitreal injection out to Week 24 Primary Endpoint
  Arms: Sham

SUMMARY:
This is a phase 3 study to determine the efficacy of VEGF Trap-Eye injected into the eye on vision function in subjects with macular edema as a consequence of central retinal vein occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects at least 18 years of age with center-involved macular edema secondary to CRVO with mean central retinal thickness ≥ 250 μm on OCT
* ETDRS best corrected visual acuity of 20/40 to 20/320 (73 to 24 letters) in the study eye

Exclusion Criteria:

* Previous treatment with anti-angiogenic drugs in the study eye (Pegaptanib sodium,anecortave acetate, bevacizumab, ranibizumab, etc.)
* Prior panretinal laser photocoagulation or macular laser photocoagulation in the study eye
* CRVO disease duration > 9 months from date of diagnosis
* Previous use of intraocular corticosteroids in the study eye or use of periocular corticosteroids in the study eye within the 3 months prior to Day 1
* Iris neovascularization, vitreous hemorrhage, traction retinal detachment, or preretinal fibrosis involving the macula in either the study eye or fellow eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2009-07; Primary Completion 2010-10 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (59):
- United States (44):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Arcadia, California
  - Beverly Hills, California
  - La Jolla, California
  - Mountain View, California
  - Oakland, California
  - Sacramento, California
  - Torrance, California
  - New London, Connecticut
  - Altamonte Springs, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Miami, Florida
  - Palm Beach Gardens, Florida
  - Winter Haven, Florida
  - Augusta, Georgia
  - Chicago, Illinois
  - Wichita, Kansas
  - Baltimore, Maryland
  - Hagerstown, Maryland
  - Towson, Maryland
  - Boston, Massachusetts
  - Grand Rapids, Michigan
  - Jackson, Michigan
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Northfield, New Jersey
  - Toms River, New Jersey
  - Rochester, New York
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Salem, Oregon
  - Kingston, Pennsylvania
  - Pittsburgh, Pennsylvania
  - West Columbia, South Carolina
  - Rapid City, South Dakota
  - Nashville, Tennessee
  - Abilene, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Antonio, Texas
- Canada (6):
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Halifax, Nova Scotia
  - London, Ontario
  - Mississauga, Ontario
  - Toronto, Ontario
- Colombia (2):
  - Medellín, Antioquia
  - Bogotá
- India (3):
  - Hyderabad, A.p.
  - Bangalore, Karnataka
  - Kolkata, West Bengal
- Israel (4):
  - Kfar Saba, Israel
  - Petah Tikva, Israel
  - Rehovot, Israel
  - Tel Aviv, Israel

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 55 study centers in the United States, Canada, Columbia, India, and Israel. The recruitment period occurred between 08 Jul 2009 and 29 Apr 2010.
Pre-assignment Details: 273 participants were screened, 189 randomized, and 188 were included in the Safety Analysis Set (SAF). The Full Analysis Set (FAS) included 187 participants with at least one post-baseline assessment.
Groups:
- Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye): Participants received a 2 mg Intravitreal Aflibercept Injection (IAI) every 4 weeks (2Q4) from Baseline (Day 1) to Week 24.
  Starting at week 24 through week 52, participants were evaluated monthly to receive either the 2 mg IAI PRN or sham injection according to the protocol re-treatment criteria as assessed by the masked physician. If none of the re-treatment criteria were met, participants received a sham injection.
  From Week 52 to 100, participants were evaluated every three months, but could receive injections of IAI up to monthly if re-treatment criteria were met; sham injections were not given. Participants were observed from Week 24 to Week 100. Participants in the safety population that completed Week 24 were at risk.
- Sham Treatment: Participants received sham treatment every 4 weeks from Baseline (Day 1) to Week 24.
  Starting at week 24 through week 52, participants were eligible for active treatment and were evaluated monthly to receive either 2 mg IAI PRN or sham injection according to the protocol re-treatment criteria as assessed by the masked physician.
  From Week 52 to 100, participants were evaluated every three months, but could receive injections of IAI up to monthly if re-treatment criteria were met; sham injections were not given.
Period: Overall Study
Arm/Group | Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) | Sham Treatment
Started | 115 | 74
Participants Received Treatment | 114 (Safety population (SAF)) | 74
Full Analysis Set (FAS) Population | 114 (FAS population used for analysis of Primary and Secondary Outcome Measures) | 73
Completed | 110 (110 Participants completed Week 24, From FAS; 102 Participants completed up to Week 100, From SAF) | 60 (60 Participants completed Week 24, From FAS; 50 Participants completed up to Week 100, From SAF)
Not Completed | 5 | 14
Not completed — Adverse Event | 0 | 3
Not completed — Death | 0 | 2
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Lack of Efficacy | 0 | 4
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye): Participants received a 2 mg Intravitreal Aflibercept Injection (IAI) every 4 weeks (2Q4) from Baseline (Day 1) to Week 24.
- Sham Treatment: Participants received sham treatment every 4 weeks from Baseline (Day 1) to Week 24.
- Total: Total of all reporting groups
Arm/Group | Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) | Sham Treatment | Total
Number analyzed (Participants) | 114 | 74 | 188
Age Continuous [Mean (Standard Deviation); unit: years] | 65.5 (13.57) | 67.5 (14.22) | 66.3 (13.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 35 | 80
  Male | 69 | 39 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 12 | 30
  Not Hispanic or Latino | 96 | 62 | 158
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 7 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 5 | 10
  White | 88 | 60 | 148
  More than one race | 12 | 6 | 18
  Unknown or Not Reported | 0 | 0 | 0
Baseline Retinal Thickness by Optical Coherence Tomography (OCT) [Mean (Standard Deviation); unit: microns] | 661.7 (237.37) | 678.4 (248.66) | 668.1 (241.23)
Baseline National Eye Institute 25-item Visual Function Questionnaire (NEI VFQ-25) Total Score [Mean (Standard Deviation); unit: scores on a scale] — The NEI VFQ-25 total score ranges from 0-100 with a score of 0 being the worst outcome and 100 being the best outcome. The NEI VFQ questionnaire is organized as a collection of subscales which are all scored from 0-100. To reach the overall composite score, each sub-scale score is averaged in order to give each sub-scale equal weight.
  scores on a scale | 77.67 (15.96) | 78.01 (16.26) | 77.81 (16.04)
Baseline Intraocular Pressure [Mean (Standard Deviation); unit: millimeters of mercury (mmHg)] | 15.1 (3.26) | 15.0 (2.83) | 15.1 (3.09)
Number of Participants with Retinal Perfusion at Baseline [Number; unit: participants] — Retinal Perfusion defined as less than 10 disc areas of capillary non-perfusion using fluorescein angiography (FA).
  Non-Perfused defined as greater than or equal to 10 disc areas of non-perfusion.
  Indeterminate defined as not able to be determined by the reading center; for the purposes of analysis, indeterminate patients were considered non-perfused.
  participants
    Perfused | 77 | 50 | 127
    Non-Perfused | 17 | 12 | 29
    Indeterminate | 20 | 12 | 32
Baseline Best Corrected Visual Acuity (BCVA) Letter Score [Mean (Standard Deviation); unit: letters correctly read] — Only participants with an ETDRS (Early Treatment Diabetic Retinopathy Study) Best Corrected Visual Acuity letter score of 73 to 25 (= Acuity of 20/40 to 20/320) in the study eye at 4 meters were included; a higher score represents better functioning.
  letters correctly read | 50.7 (13.90) | 48.7 (14.41) | 49.9 (14.10)
Time Since Central Retinal Vein Occlusion (CRVO) Diagnosis [Number; unit: participants]
  </= 2 Months | 64 | 53 | 117
  > 2 Months | 49 | 21 | 70
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Gained at Least 15 Letters in BCVA at Week 24 as Measured by ETDRS Letter Score
Description: Percentage values indicate the number of subjects in each arm who were able to read an additional 15 letters or more at Week 24 compared to baseline.
  Defined study baseline range of ETDRS Best Corrected Visual Acuity letter score of 73 to 24 letters (= Acuity of 20/40 to 20/320) in the study eye; a higher score represents better functioning.
Time Frame: Baseline and at Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) | Sham Treatment
Number analyzed (Participants) | 114 | 73
percentage of participants | 64 | 9
Statistical Analysis 1: Comparison: Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) vs Sham Treatment; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — P-value for the primary endpoint was calculated using 2-sided Cochran-Mantel-Haenszel test adjusted by regions (North America vs. Rest of World) and baseline BCVA (BCVA > 20/200 and BCVA ≤ 20/200); CMH adjusted difference; Risk Difference (RD) = 44.8, 95% CI 2-sided [33.0 to 56.6] — The Risk Difference (RD) indicates the difference between the IAI (EYLEA, VEGF Trap-Eye) Treatment group minus the Sham Treatment group

2. Secondary Outcome: Change From Baseline in BCVA as Measured by ETDRS Letter Score at Week 24 - Last Observation Carried Forward (LOCF)
Description: Defined study baseline range of ETDRS Best Corrected Visual Acuity letter score of 73 to 24 (= Acuity of 20/40 to 20/320) in the study eye; a higher score represents better functioning.
Time Frame: Baseline and at Week 24
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: letters correctly read
Arm/Group | Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) | Sham Treatment
Number analyzed (Participants) | 114 | 73
letters correctly read | 17.3 (12.78) | -4.0 (17.96)
Statistical Analysis 1: Comparison: Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) vs Sham Treatment; Test type: Superiority or Other; p < 0.0001, ANCOVA; Risk Difference (RD) = 21.70, 95% CI 2-sided [17.36 to 26.04] — RD is the IAI group minus sham group. 95% confidence interval is for the RD
Statistical Analysis 2: Comparison: Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) vs Sham Treatment; Test type: Superiority or Other; ANCOVA; Least Square Mean = 16.36 — LS Mean indicates is the IAI (EYLEA, VEGF Trap-Eye) Treatment group minus the Sham Treatment group

3. Secondary Outcome: Change From Baseline in Central Retinal Thickness (CRT) at Week 24 - LOCF
Time Frame: Baseline and at Week 24
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) | Sham Treatment
Number analyzed (Participants) | 114 | 73
microns | -457.2 (238.21) | -144.8 (291.07)
Statistical Analysis 1: Comparison: Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) vs Sham Treatment; Test type: Superiority or Other; p < 0.0001, ANCOVA; Risk Difference (RD) = -311.9, 95% CI 2-sided [-389.4 to -234.4] — The Risk Difference (RD) indicates the difference between the IAI (EYLEA, VEGF Trap-Eye) Treatment group minus the Sham Treatment group. 95% confidence interval is for the RD
Statistical Analysis 2: Comparison: Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) vs Sham Treatment; Test type: Superiority or Other; ANCOVA; Least Square Mean = -487.1 — The Least Square Mean indicates the difference between the IAI (EYLEA, VEGF Trap-Eye) Treatment group minus the Sham Treatment group

4. Secondary Outcome: Percentage of Participants Progressing to Any of the Following: Anterior Segment Neovascularization, New Vessels of the Disc (NVD) or New Vessels Elsewhere (NVE) During the First 24 Weeks
Time Frame: Baseline to Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) | Sham Treatment
Number analyzed (Participants) | 114 | 73
percentage of participants
  Any neovascularization | 0 | 6.8
  Anterior segment neovascularization | 0 | 6.8
  Neovascularization of the optic disc (NVD) | 0 | 0
  Neovascularization elsewhere in the fundus (NVE) | 0 | 0
Statistical Analysis 1: Comparison: Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) vs Sham Treatment; Test type: Superiority or Other; p = 0.0059, Cochran-Mantel-Haenszel; CMH adjusted difference; Risk Difference (RD) = -6.6, 95% CI 2-sided [-12.2 to -1.1] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Change From Baseline in the NEI VFQ-25 in Total Score at Week 24 (LOCF)
Description: The NEI VFQ-25 assesses visual function and quality of life. Total score ranges from 0-100 with a score of 0 being the worst outcome and 100 being the best outcome. The NEI VFQ questionnaire is organized as a collection of subscales which are all scored from 0-100. To reach the overall composite score, each sub-scale score is averaged in order to give each sub-scale equal weight.
Time Frame: Baseline and at Week 24
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) | Sham Treatment
Number analyzed (Participants) | 114 | 73
scores on a scale | 7.2 (12.11) | 0.8 (9.79)
Statistical Analysis 1: Comparison: Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) vs Sham Treatment; Test type: Superiority or Other; p = 0.0009, ANCOVA; Risk Difference (RD) = 6.26, 95% CI 2-sided [2.61 to 9.91] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) vs Sham Treatment; Test type: Superiority or Other; ANCOVA; Least Square Mean = 8.80 — Least Square Mean indicates the difference between the IAI (EYLEA, VEGF Trap-Eye) Treatment group minus the Sham Treatment group

ADVERSE EVENTS:
Time Frame: Baseline to Week 24; Week 24 to Week 100
Description: Adverse event data were collected from the sites during the time period from Baseline through Week 24 or/and Week 100. For analysis, adverse events with a start date on or after the Week 24 visit date are summarized in the Week 24 to Week 100 time period.
Groups:
- Intravitreal Aflibercept Injection (IAI) (Baseline to Week 24): Participants received a 2 mg Intravitreal Aflibercept Injection (IAI) every 4 weeks (2Q4) from Baseline (Day 1) to Week 20. Participants were observed until Week 24.
  Participants in the safety population were at risk.
- Sham Treatment (Baseline to Week 24): Participants received sham treatment every 4 weeks from Baseline (Day 1) to Week 20. Participants were observed until Week 24. Participants in the safety population were at risk.
- IAI to IAI (Week 24 to Week 100): Starting at week 24 through week 52, participants were evaluated monthly to receive either the 2 mg Intravitreal Aflibercept Injection (IAI) PRN or sham injection according to the protocol re-treatment criteria as assessed by the masked physician. If none of the re-treatment criteria were met, participants received a sham injection.
  From Week 52 to 100, participants were evaluated every three months, but could receive injections of IAI up to monthly if re-treatment criteria were met; sham injections were not given. Participants were observed from Week 24 to Week 100. Participants in the safety population that completed Week 24 were at risk.
- Sham Treatment to IAI (Week 24 to Week 100): Starting at week 24 through week 52, participants were eligible for active treatment and were evaluated monthly to receive either 2 mg Intravitreal Aflibercept Injection (IAI) PRN or sham injection according to the protocol re-treatment criteria as assessed by the masked physician.
  From Week 52 to 100, participants were evaluated every three months, but could receive injections of IAI up to monthly if re-treatment criteria were met; sham injections were not given.
Arm/Group | Intravitreal Aflibercept Injection (IAI) (Baseline to Week 24) | Sham Treatment (Baseline to Week 24) | IAI to IAI (Week 24 to Week 100) | Sham Treatment to IAI (Week 24 to Week 100)
Serious Adverse Events (participants affected / at risk) | 6/114 | 6/74 | 20/110 | 14/60
Other Adverse Events (participants affected / at risk) | 57/114 | 34/74 | 76/110 | 50/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intravitreal Aflibercept Injection (IAI) (Baseline to Week 24) (N=114) | Sham Treatment (Baseline to Week 24) (N=74) | IAI to IAI (Week 24 to Week 100) (N=110) | Sham Treatment to IAI (Week 24 to Week 100) (N=60)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Pernicious anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Oesophageal adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 — Ocular AE Fellow Eye
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 — Ocular AE Fellow Eye
Cystoid macular oedema (Eye disorders) | 0 | 0 | 2 | 0 — Ocular AE Study Eye
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 — Ocular AE Study Eye
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 — Ocular AE Study Eye
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 — Ocular AE Study Eye
Glaucoma (Eye disorders) | 0 | 2 | 0 | 1 — Ocular AE Study Eye
Iris neovascularisation (Eye disorders) | 0 | 2 | 0 | 0 — Ocular AE Study Eye
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 — Ocular AE Study Eye
Macular fibrosis (Eye disorders) | 0 | 0 | 1 | 0 — Ocular AE Fellow Eye
Macular oedema (Eye disorders) | 0 | 0 | 1 | 0 — Ocular AE Study Eye
Maculopathy (Eye disorders) | 0 | 0 | 0 | 0 — Ocular AE Study Eye
Optic disc vascular disorder (Eye disorders) | 0 | 0 | 0 | 0 — Ocular AE Study Eye
Posterior capsule opacification (Eye disorders) | 0 | 0 | 1 | 0 — Ocular AE Fellow Eye
Retinal artery occlusion (Eye disorders) | 1 | 0 | 0 | 0 — Ocular AE Study Eye
Retinal exudates (Eye disorders) | 0 | 0 | 0 | 0 — Ocular AE Study Eye
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 — Ocular AE Fellow Eye
Retinal pigment epitheliopathy (Eye disorders) | 0 | 0 | 0 | 0 — Ocular AE Study Eye
Retinal tear (Eye disorders) | 0 | 1 | 0 | 1 — Ocular AE Study Eye
Retinal vascular disorder (Eye disorders) | 0 | 0 | 1 | 0 — Ocular AE Study Eye
Retinal vein occlusion (Eye disorders) | 0 | 1 | 1 | 0 — Ocular AE Study Eye
Visual acuity reduced (Eye disorders) | 1 | 1 | 1 | 0 — Ocular AE Study Eye
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 0 — Ocular AE Study Eye
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 — Ocular AE Study Eye
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 — Ocular AE Fellow Eye
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Adhesion (General disorders) | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 2 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis viral (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 0
Clostridial infection (Infections and infestations) | 0 | 1 | 0 | 0
Endophthalmitis (Infections and infestations) | 1 | 0 | 0 | 0 — Ocular AE Study Eye
Herpes oesophagitis (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 — Ocular AE Fellow Eye
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 — Ocular AE Study Eye
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 — Ocular AE Fellow Eye
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Renal haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood pressure systolic increased (Investigations) | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 0 | 0 | 1 | 0 — Ocular AE Fellow Eye
Protein urine present (Investigations) | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 2
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Dementia (Nervous system disorders) | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intravitreal Aflibercept Injection (IAI) (Baseline to Week 24) (N=114) | Sham Treatment (Baseline to Week 24) (N=74) | IAI to IAI (Week 24 to Week 100) (N=110) | Sham Treatment to IAI (Week 24 to Week 100) (N=60)
Hypertension (Vascular disorders) | 10 | 4 | 13 | 9
Cataract (Eye disorders) | 0 | 0 | 6 | 0 — Ocular AE Fellow Eye
Cystoid macular oedema (Eye disorders) | 0 | 0 | 14 | 4 — Ocular AE Study Eye
Dry eye (Eye disorders) | 0 | 0 | 0 | 4 — Ocular AE Study Eye
Eye irritation (Eye disorders) | 6 | 0 | 0 | 0 — Ocular AE Study Eye
Eye pain (Eye disorders) | 16 | 4 | 9 | 4 — Ocular AE Study Eye
Iris neovascularisation (Eye disorders) | 0 | 4 | 0 | 0 — Ocular AE Study Eye
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 4 — Ocular AE Study Eye
Macular oedema (Eye disorders) | 0 | 0 | 20 | 0 — Ocular AE Study Eye
Maculopathy (Eye disorders) | 10 | 0 | 6 | 0 — Ocular AE Study Eye
Optic disc vascular disorder (Eye disorders) | 8 | 0 | 6 | 5 — Ocular AE Study Eye
Retinal exudates (Eye disorders) | 7 | 0 | 0 | 5 — Ocular AE Study Eye
Retinal haemorrhage (Eye disorders) | 0 | 0 | 6 | 4 — Ocular AE Fellow Eye
Retinal pigment epitheliopathy (Eye disorders) | 0 | 0 | 0 | 12 — Ocular AE Study Eye
Retinal vascular disorder (Eye disorders) | 6 | 4 | 8 | 0 — Ocular AE Study Eye
Visual acuity reduced (Eye disorders) | 7 | 12 | 27 | 8 — Ocular AE Study Eye
Vitreous detachment (Eye disorders) | 0 | 5 | 8 | 0 — Ocular AE Study Eye
Vitreous floaters (Eye disorders) | 6 | 0 | 0 | 0 — Ocular AE Study Eye
Influenza (Infections and infestations) | 0 | 0 | 7 | 0
Nasopharyngitis (Infections and infestations) | 0 | 4 | 6 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 0 | 6 | 0
Blood pressure systolic increased (Investigations) | 0 | 0 | 0 | 4
Blood urine present (Investigations) | 0 | 0 | 0 | 4
Intraocular pressure increased (Investigations) | 0 | 0 | 0 | 4 — Ocular AE Fellow Eye
Protein urine present (Investigations) | 0 | 0 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI, after completion of the trial and multi-center publication, is that the sponsor can review results communications prior to public release & may have the right to embargo communications regarding results for a period between 60 & 180 days from the time submitted to the sponsor for review; provided that the sponsor can remove confidential/proprietary information. The sponsor cannot require other changes to the communication and cannot extend the embargo.